CLINICAL TRIAL: NCT07086833
Title: The Food Environment, Microbial Cysteine Metabolism, and Cancer Disparities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: American Cancer Society, Inc. (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Patricia Wolf, Dr. Patricia Wolf, Assistant Professor, Department of Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-2023-1426; RSG-23-1154989-01-CSCT (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Risk; Colorectal Cancer Prevention; Colorectal Cancer; Diet Modification; Dietary Intervention; Cancer Prevention
Keywords: Intestinal Neoplasms; Neoplasms; Colonic Diseases; Colorectal Cancer; Colorectal Neoplasms; Gut Microbiome; Cysteine Metabolism; Colorectal Adenomas; Intestinal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Neoplasms; Colonic Diseases; Intestinal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled cross-over feeding trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High cysteine diet (Experimental): Participants will eat a diet higher in cysteine, relying on more animal based protein.
  Interventions: Other: High Cysteine Diet
- Low cysteine diet (Experimental): Participants will eat a diet lower in cysteine, relying on more plant based protein.
  Interventions: Other: Low Cysteine Diet

INTERVENTIONS:
Other: Low Cysteine Diet — A diet low in cysteine, about 1.4 g/1000 kcal.
  Arms: Low cysteine diet
Other: High Cysteine Diet — A diet high in cysteine, about 3 g/1000 kcal.
  Arms: High cysteine diet

SUMMARY:
The goal of this clinical trial is to learn if changing cysteine levels in the diet can influence how the body processes cysteine in Black and White individuals aged 45-75 with a history of non-cancerous polyps. The main questions it aims to answer are:

* At the beginning of the study, do Black participants have higher levels of cortisol (a stress hormone) and compounds made from cysteine in their blood when compared to White participants?
* Does eating less cysteine lower the body's natural cysteine activity and lead to less gut bacteria that break down cysteine?
* Does eating less cysteine lead to less inflammation in the gut and lower levels of markers of inflammation in the blood?

Research will compare a high cysteine diet and a low cysteine diet, and each participant will eat both diets.

Participants will be in the study for 11 weeks and 2 days. Over the course of the study, participants will:

* Eat a high cysteine diet for 3 weeks, and a low cysteine diet for 3 weeks
* Eat a moderate cysteine diet for 1 week before each study diet
* Complete surveys
* Provide blood, stool, and saliva samples
* Maintain food logs

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-75
* Up to date with CRC screening colonoscopy with a high risk of CRC, defined as a history of 3 or more adenomatous polyps (APs) or an AP >1 cm in the past 5 years
* Identify as Black or Non-Hispanic White
* If female, no menstrual period for at least six months
* Willingness to donate oral wash and stool samples
* Willingness to complete 24-hour dietary recalls

Exclusion Criteria:

* Antibiotic use within the last 6 months
* Abnormal gastrointestinal transit
* A history of organ transplantation
* Use of illicit drugs, combustible tobacco, or dietary supplements
* Pre- or probiotics within the last two months
* A history of cancer treatment within the past 12 months
* CRC or a genetic predisposition to CRC
* A baseline body weight > 450 lbs
* Weight gain or loss > 4 kg 3 months prior to study
* Significant food allergies, food preferences or therapeutic or vegetarian diets
* Menstrual cycle within the last 6 months
* Antibiotics in the last 2 months
* Cannot keep a food record for 7 consecutive days during screening after detailed instruction
* Significant medical conditions
* History of eating disorders
* Alcoholism
* Individuals under the age of 18

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Colonic inflammation | Baseline, Week 1 (Day 8), Week 2 (Day 15), Week 4 (Day 29), Week 7 (Day 49), Week 8 (Day 57), Week 9 (Day 64), Week 11 (Day 78)
  Fecal calprotectin, a marker of intestinal inflammation, will be measured from 100 mg of stool collected at the respective timeframe using a CALPRO Calprotectin ELISA test.
Fecal microbial content | Baseline, Week 1 (Day 8), Week 2 (Day 15), Week 4 (Day 29), Week 7 (Day 49), Week 8 (Day 57), Week 9 (Day 64), Week 11 (Day 78)
  Microbial genomic DNA will be extracted from stool obtained at the respective timeframe using a Qiagen DNeasy PowerSoil Kit. Genomic DNA will be fragmented using a Covaris S2 and processed into libraries using an Integrated DNA Technologies xGen DNA Library Prep Kit. Final libraries will be pooled and sequenced on an Illumina NovaSeq X using 25B chemistry.
Systemic markers of inflammation | Baseline, Week 1 (Day 9), Week 2 (Day 16), Week 3 (Day 23), Week 4 (Day 30), Week 7 (Day 50), Week 8 (Day 58), Week 9 (Day 65), Week 11 (Day 79)
  Serum from blood collected at the respective timeframe will be analyzed in triplicate with the Bio-Plex® Precision Pro™ (Bio rad, Hercules, CA) human cytokine 10-plex immunoassay to detect IL-1β, IL-6, IFN-γ, TNF-α, IL-2, IL-4, IL-5, IL-10, IL-12 (p70) and IL-13.

SECONDARY OUTCOMES:
Quantification of serum hydroxycortisol and cysteine metabolism markers | Baseline, Week 1 (Day 9), Week 2 (Day 16), Week 3 (Day 23), Week 4 (Day 30), Week 7 (Day 50), Week 8 (Day 58), Week 9 (Day 65), Week 11 (Day 79)
  Serum hydroxycortisol and measures of cysteine metabolism (cysteine, homocysteine, lanthionine, cystathionine, serine) will be determined using hydrophilic interaction liquid chromatography with triple quadrupole tandem mass spectrometry by the Purdue Metabolite Profiling Facility.
Absolute and relative quantification of microbial cysteine metabolic genes | Baseline, Week 1 (Day 8), Week 2 (Day 15), Week 4 (Day 29), Week 7 (Day 49), Week 8 (Day 57), Week 9 (Day 64), Week 11 (Day 78)
  Microbial genomic DNA will be extracted from stool obtained at the respective timeframe using a Qiagen DNeasy PowerSoil Kit. To estimate gene content, metagenomic libraries will be constructed from stool DNA. Metagenomic data will be processed to filter potential host DNA sequences and remove low-quality reads. Raw shotgun data will be assembled using MEGAHIT and assembled contigs will be binned using MetaBAT2. Taxonomic classification of binned contigs will be performed using CAT/BAT and differences genera that have functional genes for sulfur metabolism will be assessed. Assembled and binned metagenomes will be surveyed for genes for cysteine metabolism using custom hidden Markov model (HMM) libraries.
Whole body composition | Baseline, Week 4 (Day 30), Week 11 (Day 79)
  DXA whole-body composition scan
Exfoliated intestinal epithelial cell transcriptomics | Baseline, Week 1 (Day 8), Week 4 (Day 29), Week 8 (Day 57), Week 11 (Day 78)
  Exfoliated intestinal epithelial cells separated from stool collected at the respective timeframe with gene expression analysis

OTHER OUTCOMES:
Psychosocial health | Baseline, Week 4 (Day 30), Week 8 (Day 58),Week 11 (Day 79)
  survey
Medication use | Baseline, Week 4 (Day 30), Week 8 (Day 58),Week 11 (Day 79)
  survey
Bowel habits | Baseline, Week 4 (Day 30), Week 8 (Day 58),Week 11 (Day 79)
  survey

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Hospital Clinical Research Center, Indianapolis, Indiana
  - Purdue Clinical Research Center, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: No